CLINICAL TRIAL: NCT04532112
Title: Biocontainment Device With Aerosol Clearance for Aerosol Generating Procedures
Brief Title: Biocontainment Device for Aerosol Generating Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 843373
Record Dates: First submitted 2020-08-13; First posted 2020-08-31 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Protective Device (Physical Object); Aerosol Disease; Droplet Spread
Keywords: PPE-personal protective equipment

STUDY DESIGN:
Intervention Model Description: The intervention consists of a biocontainment and aerosol clearance device that will be tested in the controlled setting to assess feasibility to perform airway procedures under general anesthesia with the device. There is no specific control device for this product. The control condition for this intervention will consist of airway procedures per routine clinical protocols without the biocontainment device. This study will be performed initially in locations where a patient would undergo a scheduled airway procedure under general anesthesia on non-COVID-19 patients. All participants in this study as well as non-participants who are present in the room during the airway procedure (aerosol-generating procedure) will continue to use appropriate level of PPE per hospital protocols and policies. This device does not replace standard aerosol-protecting PPE.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intubated Subjects with the Biocontainment Device (Experimental): Subjects undergoing scheduled airway procedures under general anesthesia with the Biocontainment Device by anesthesiologists trained in device use.
  Interventions: Device: Biocontainment Device For Aerosol Generating Procedures (Biobox)
- Intubated Subjects without the Biocontainment Device (Placebo Comparator): Subjects undergoing scheduled airway procedures under general anesthesia with the Biocontainment Device by same cohort of anesthesiologists trained in device use.
  Interventions: Device: Control for aerosol generating procedures

INTERVENTIONS:
Device: Biocontainment Device For Aerosol Generating Procedures (Biobox) — The intervention consists of a biocontainment and aerosol evacuation device (Biobox) that will be placed around a patient prior to the airway procedure and remain in place throughout the airway procedure. The Biobox device is manufactured by National Flag and consists of a re-useable frame with a disposable, plastic torso drape. This is a new device that has not been used previously in a healthcare setting.
  Arms: Intubated Subjects with the Biocontainment Device
Device: Control for aerosol generating procedures — There is no control device for the aerosol containment device. As such, intubation without a device will serve as the control/placebo arm for this trial.
  Arms: Intubated Subjects without the Biocontainment Device

SUMMARY:
The primary goal of this study is to assess use of a biocontainment device for planned airway procedures under general anesthesia. This will serve as a platform for using this device as a novel biocontainment and aerosol evacuation system as part of rapid sequence intubation protocols for COVID-19 patients. We hypothesize that airway procedures with the aerosol biocontainment device will be safe and effective with airway procedure times approaching times for airway procedures without the device.

DETAILED DESCRIPTION:
This is a multi-site (two sites), unblinded, randomized, observational study performed in a controlled environment in the operating room. The hypothesis is that rapid sequence intubation or other urgent airway procedures performed with the biocontainment device will be safe and can be performed in an equivalent manner to urgent airway procedures without the biocontainment device. Methods to minimize bias include randomizing patients to intubation with or without the biocontainment device.

ELIGIBILITY:
Inclusion Criteria:

A) User (healthcare worker):

• Anesthesiologist, anesthesia resident, or CRNA at the Hospital of the University of Pennsylvania or PPMC who has signed and dated informed consent.

B) Patient:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* ASA I, II, III
* Undergoing planned procedure involving an airway procedure under general anesthesia

Exclusion Criteria:

A) User (healthcare worker):

• Pregnancy due to potential risks from lifting the device.

B) Patient:

* Known history of difficult airway
* Anticipated difficult airway management for any reason
* COVID-19 positive status
* Pregnancy
* Planned prolonged intubation post-surgery or anticipated inability to answer patient questionnaire within 1 week of intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Atkins, Md, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intubated Subjects Without the Biocontainment Device: Subjects undergoing scheduled airway procedures under general anesthesia with the Biocontainment Device by anesthesiologists trained in device use.
  Control for aerosol generating procedures: There is no control device for the aerosol containment device. As such, intubation without a device will serve as the control/placebo arm for this trial.
Period: Overall Study
Arm/Group | Intubated Subjects With the Biocontainment Device | Intubated Subjects Without the Biocontainment Device
Started | 25 | 12
Completed | 22 | 12
Not Completed | 3 | 0
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intubated Subjects With the Biocontainment Device | Intubated Subjects Without the Biocontainment Device | Total
Number analyzed (Participants) | 25 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (16.8) | 56 (9.1) | 53.7 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 8 | 25
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 22 | 11 | 33
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 19 | 8 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 12 | 37
chronic lung disease or moderate/severe asthma [Count of Participants; unit: Participants] | 3 | 2 | 5
cardiac disease [Count of Participants; unit: Participants] | 8 | 3 | 11
obstructive sleep apnea [Count of Participants; unit: Participants] | 4 | 1 | 5
diabetes [Count of Participants; unit: Participants] | 1 | 1 | 2
immunocompromised [Count of Participants; unit: Participants] | 0 | 1 | 1
ASA status [Count of Participants; unit: Participants] — ASA status is the American Society of Anesthesiologists status for screening overall patient health in the context of a planned surgical procedure. Grading is as noted below ASA I: A normal healthy patient ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life
  Participants
    ASA II | 17 | 8 | 25
    ASA III | 8 | 4 | 12
Mallampati [Count of Participants; unit: Participants] — Mallampati score describes the size of the tongue base relative to oropharynx opening to characterize the amount of open space in the oropharynx. A grade of I is considered a wide open airway and a grade of IV is considered a crowded airway that is more likely to have airway obstruction.
  Participants
    Mallampati 1 | 8 | 3 | 11
    Mallampati 2 | 12 | 5 | 17
    Mallampati 3 | 5 | 4 | 9
    Mallampati 4 | 0 | 0 | 0
BMI [Count of Participants; unit: Participants]
  <20 | 0 | 3 | 3
  20-24.99 | 7 | 3 | 10
  25-29.99 | 11 | 2 | 13
  30-34.99 | 2 | 2 | 4
  35-39.99 | 3 | 1 | 4
  40-44.99 | 2 | 1 | 3
  >45 | 0 | 0 | 0
hyomental distance [Count of Participants; unit: Participants]
  normal | 24 | 11 | 35
  short | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Measuring the Time for Performing an Airway Procedure With or Without the Biocontainment Device.
Description: Measure the amount of time it take to perform an airway procedure (intubation) with or without the biocontainment device.
Time Frame: Start of airway procedure through to completion of airway procedure.
Measure: Median (Standard Deviation); unit: time (seconds)
Arm/Group | Intubated Subjects With the Biocontainment Device | Intubated Subjects Without the Biocontainment Device
Number analyzed (Participants) | 22 | 12
time (seconds) | 46 (26.9) | 37 (13.1)

2. Primary Outcome: Quantifying the Number of AEs or ADEs to Assess Device Safety.
Description: Measure the number of adverse events, adverse device events associated with using the biocontainment device.
Time Frame: collected at time of procedure, on average within 3 minutes of starting the procedure
Measure: Number; unit: number of events
Arm/Group | Intubated Subjects With the Biocontainment Device | Intubated Subjects Without the Biocontainment Device
Number analyzed (Participants) | 25 | 12
number of events | 3 | 0

3. Secondary Outcome: Median Likert Ratings From Device Use Survey Questions That Assess User Subject Device Comfort.
Description: Assess the user subject's comfort with using the biocontainment device. 5 point Likert scale (1. Strongly disagree, 2. disagree, 3. neutral, 4. agree, 5. strongly agree). data shown is median score of participants. A higher score would mean a better outcome.
Time Frame: Survey completed up to 1 day after airway procedure
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Intubated Subjects With the Biocontainment Device
Number analyzed (Participants) | 25
score on a scale | 3 (0.77)

4. Secondary Outcome: Median Likert Ratings From Device Use Survey Questions That Assess User Subject Healthcare Burden With the Device.
Description: Assess for additional healthcare and cognitive burden imposed by the device. 5 point Likert scale (1. Strongly disagree, 2. disagree, 3. neutral, 4. agree, 5. strongly agree). data shown is median score of participants. A higher score would mean a worse outcome.
Time Frame: Survey completed up to 1 day after completion of airway procedure
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Intubated Subjects With the Biocontainment Device
Number analyzed (Participants) | 25
score on a scale | 4 (0.84)

5. Secondary Outcome: Median Likert Rating of the Patient Questionnaire Results to Assess Patient Experience in the Device.
Description: Survey of patient's post-procedure on experience being inside the device. 5 point Likert scale (1. Strongly disagree, 2. disagree, 3. neutral, 4. agree, 5. strongly agree). data shown is median score of participants. A higher score means a better outcome.
Time Frame: Survey completed up to 1 day after airway procedure
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Intubated Subjects With the Biocontainment Device
Number analyzed (Participants) | 20
score on a scale | 4 (0.87)

ADVERSE EVENTS:
Time Frame: adverse events were collected at the time of the procedure, on average within 3 minutes of starting the procedure.
Arm/Group | Intubated Subjects With the Biocontainment Device | Intubated Subjects Without the Biocontainment Device
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/12
Other Adverse Events (participants affected / at risk) | 3/25 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intubated Subjects With the Biocontainment Device (N=25) | Intubated Subjects Without the Biocontainment Device (N=12)
expected adverse event (Surgical and medical procedures) | 1 (1) | 0 (0) — device removed due to subject anxiety and claustrophobia
expected adverse event (Surgical and medical procedures) | 2 (2) | 0 (0) — difficult intubation. device removed to successfully perform intubation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT04532112/Prot_SAP_000.pdf